CLINICAL TRIAL: NCT01607047
Title: Utility of Quantitative Polymerase Chain Reaction to Predict Clinical Outcome of Leptospirosis in French West Indies
Brief Title: French West Indies Leptospirosis Study
Acronym: LEPTO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: Clinique Antilles-Guyane (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHU FDF 10/B/13
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Leptospirosis
Keywords: leptospirosis; qPCR; cohort; french west indies; blood sample collection; pronostic; diagnosis
MeSH Terms: conditions — Leptospirosis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, plasma, DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
Leptospirosis is a zoonosis of worldwide distribution whose incidence is higher in the tropics, where conditions for transmissions are favorable. The disease is endemic in Martinique and Guadeloupe, two Caribbean islands of the French West Indies. In tropical areas, many wild and domestic animals serve as reservoirs for pathogenic Leptospira strains and contaminate the environment by shedding the organisms in their urine. Humans are usually infected through abraded skin or mucous membrane contact with water contaminated by the urine of animal reservoirs, and less frequently by direct contact with animals or their urine. The mean incubation period is 10 days, with a usual range of 2-20 days. Clinical manifestations are protean and the spectrum of symptoms range from subclinical or mild anicteric febrile illness to acute renal failure and respiratory distress syndrome which are associated with high mortality rates.

The microscopic agglutination test (MAT) and culture are the reference standard test for diagnosis of leptospirosis, but they are only available in reference laboratories and their conclusive results requires convalescent sample or prolonged incubation. At present, only direct detection methods using PCR might provide rapid diagnosis during the early acute stage of the illness, when treatment is likely to have the greatest benefit.

Quantitative PCR also offers the ability to measure level of leptospiremia in clinical samples. Using qPCR based diagnosis, the investigators have the opportunity to study the association of level of leptospiremia and clinical manifestations in French West Indies. All qPCR-positive samples will be used for molecular typing.

DETAILED DESCRIPTION:
Principal objective

To determine if leptospiral bacterial load is associated with severe evolution of the disease (organ failure, internal bleeding, death) in French West Indies.

Secondary objective

1. To identify demographic, clinical, biological, bacteriological, and genetic factors (HLA) associated with severe complications of leptospirosis (organ failure, internal bleeding, death).
2. To identify demographic, clinical, biological, bacteriological, and genetic factors (HLA) associated with an altered quality of life after the acute phase of leptospirosis.
3. To collect human biological samples to allow studies of the individual susceptibility to the infection (genetic polymorphisms, HLA).

ELIGIBILITY:
Inclusion Criteria:

* Adults (more than 18 years)
* Consulting a participating hospital center (emergency room, full hospitalization, day hospitalization, or outpatient visit).
* Diagnosis of leptospirosis confirmed by qPCR
* Possibility of follow-up throughout the 12-week study period.
* Patient registered in the French medical social security national program
* Acceptance to participate in the study and in follow-up; informed consent of the patient or a legal representative (patients unable to sign the consent form).

Exclusion Criteria:

* Negativity of leptospirosis qPCR based diagnosis
* Children under 18 years old
* No possible follow-up after the first visit
* Refusal to participate in the study
* Patient not registered in the French medical social security national program

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a leptospirosis diagnosis confirmed by qPCR
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-12; Primary Completion 2012-09 (Actual); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Complicated forms of leptospirosis | 12 weeks
  Occurrence, during follow-up (for 12 weeks following symptom onset), of shock, internal bleeding, failure of one or several organs or systems (brain, heart, lung, liver, kidney, clotting system), or death.

SECONDARY OUTCOMES:
quality of life | 12 weeks
  Changes in quality of life, measured with the EuroQol® questionnaire in the first 3 weeks and 12 weeks after the onset of dengue fever symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Hochedez, MD, Principal Investigator — CHU fort de france
Locations (2):
- France (2):
  - CHU Pointe-à-Pitre Abymes, Pointe à Pitre, Guadeloupe
  - CHU Martinique, Fort de France, Martinique